CLINICAL TRIAL: NCT03038217
Title: Investigation of the Value of ctDNA Analysis in the Diagnosis, Treatment, and Surveillance of Patients With Surgically Resectable Colorectal Cancer
Brief Title: Investigation of the Value of ctDNA in Diagnosis, Treatment, and Surveillance of Surgically Resectable Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Guole Lin, Professor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUMCH-Colorectal Surgery
Record Dates: First submitted 2016-12-20; First posted 2017-01-31 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Rectal Cancer, Adenocarcinoma; Neoadjuvant Chemoradiation
Keywords: rectal cancer; neoajuvant chemoradiation; circulating tumor DNA
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX; Mastectomy, Segmental

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ACT group (Experimental): Group of patients with pathologically confirmed Stage II-III colorectal cancer who receive postoperative treatment with chemotherapeutic agent (ACT) using Capecitabine +/- Oxaliplatin.
  Interventions: Drug: Capecitabine +/- Oxaliplatin
- Non-ACT group (Experimental): Group of patients with pathologically confirmed stage II colorectal cancer who receive no adjuvant chemotherapy.
  Interventions: Other: No adjuvant chemotherapy
- LR group (Experimental): Group of patients with clinically staged T1-2N0 rectal cancer who undergo local resection (LR)
  Interventions: Procedure: local resection
- RR group (Experimental): Group of patients with clinically staged T1-2N0 rectal cancer who undergo radical resection (RR)
  Interventions: Procedure: radical resection

INTERVENTIONS:
Drug: Capecitabine +/- Oxaliplatin — Patients in ACT group will undergo postoperative adjuvant chemotherapy with single agent Capecitabine regimen or combined Capecitabine +Oxaliplatin regimen.
  Arms: ACT group
Procedure: local resection — Patients in the LR group will undergo local resection of the T1-2N0 rectal carcinoma
  Other Names: LR
  Arms: LR group
Procedure: radical resection — Patients in the RR group will undergo radical resection of the T1-2N0 rectal carcinoma
  Other Names: RR
  Arms: RR group
Other: No adjuvant chemotherapy — Patients in Non-ACT group will not undergo postoperative adjuvant chemotherapy.
  Arms: Non-ACT group

SUMMARY:
In this study, we aim to investigate the value of circulating tumor DNA (ctDNA) analysis in the diagnosis, treatment, and surveillance of patients with surgically resectable colorectal cancer, by performing serial analysis of ctDNA, next-generation sequencing of surgical specimens, and observation of patients undergoing radical resection of the tumor with or without adjuvant chemo- and/or radiotherapy.

DETAILED DESCRIPTION:
A prospective, observational study to determine the value of circulating tumor DNA (ctDNA) for predicting the therapeutic effects of the combined modality treatment for colorectal cancer and the patients' long-term prognosis.

Research objects: patients with surgically resectable colorectal cancer. After giving fully informed consent, the prospective participants will undergo the classical combined modality treatment according to NCCN guidelines. Serial analysis of ctDNA will be performed at specific time points including pre-treatment, (post-NCRT for NCRT patients), postoperative week 1, post-ACT, postoperative year 1, 2, and 3. The next-generation sequencing of surgical specimens will be performed as well. Participants will be observed and examined during the entire course of treatment and the follow-up period. The 3 year disease free survival (3y-DFS) will be the primary end-point.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years old.
2. Patients with surgically resectable colorectal cancer, while without distal metastasis of the disease.
3. Patients with ASA physical status scroe of I to III.
4. Patients who can fully understand the content of the informed consent form and sign it upon their own opinions.
5. Patients who can coordinate with the researchers to undergo the long-term post-treatment rechecks and follow-ups.

Exclusion Criteria:

1. Patient has any underlying or current medical condition, which, in the opinion of the Investigator, would interfere with the evaluation of the patient (e.g., end-stage liver disease, pulmonary hypertension, systemic lupus erythematosis etc.).
2. Patient is pregnant or lactating.
3. Patient has a history of malignancy within 5 years except curatively treated basal cell carcinoma, squamous cell carcinoma in a non-mucosal, ultraviolet exposed area, or cervical carcinoma.
4. Patient is participating in any other clinical trials within 30 days prior to screening.
5. Patient has severe mental illness.
6. Patient has any other conditions, which, in the opinion of the Investigator, would interfere with the evaluation of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
5y DFS | 5 years
  The 5-year disease free survival rate of the patients.
5y LR | 5 years
  The 5-year local recurrence rate of the patients.
5y OS | 5 years
  The 5-year overall survival rate of the patients.

SECONDARY OUTCOMES:
Changes of ctDNA level after surgery | 1 month
  Changes of patients' ctDNA level after undergoing surgical resection of the tumor.
Changes of ctDNA level after adjuvant therapy | 6 months
  Changes of patients' ctDNA level after receiving adjuvant therapy (eg. adjuvant chemothearpy).
Changes of ctDNA level when disease recurs | 5 year
  Changes of patients' ctDNA level after disease recurrence happens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reinert T, Scholer LV, Thomsen R, Tobiasen H, Vang S, Nordentoft I, Lamy P, Kannerup AS, Mortensen FV, Stribolt K, Hamilton-Dutoit S, Nielsen HJ, Laurberg S, Pallisgaard N, Pedersen JS, Orntoft TF, Andersen CL. Analysis of circulating tumour DNA to monitor disease burden following colorectal cancer surgery. Gut. 2016 Apr;65(4):625-34. doi: 10.1136/gutjnl-2014-308859. Epub 2015 Feb 4. PMID 25654990
- [Background] Stroun M, Anker P, Maurice P, Lyautey J, Lederrey C, Beljanski M. Neoplastic characteristics of the DNA found in the plasma of cancer patients. Oncology. 1989;46(5):318-22. doi: 10.1159/000226740. PMID 2779946
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Background] Zhou J, Chang L, Guan Y, Yang L, Xia X, Cui L, Yi X, Lin G. Application of Circulating Tumor DNA as a Non-Invasive Tool for Monitoring the Progression of Colorectal Cancer. PLoS One. 2016 Jul 26;11(7):e0159708. doi: 10.1371/journal.pone.0159708. eCollection 2016. PMID 27459628